CLINICAL TRIAL: NCT05191017
Title: Phase 1b/2 Safety and Efficacy Study of NUV-422 in Combination With Enzalutamide in Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: Study of NUV-422 in Combination With Enzalutamide in Patients With mCRPC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Nuvation Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NUV-422-04
Record Dates: First submitted 2021-12-22; First posted 2022-01-13 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer; Prostatic Cancer; Cancer of Prostate; Cancer of the Prostate; Prostate Neoplasm; Castrate Resistant Prostate Cancer; Castration Resistant Prostatic Cancer; Castration Resistant Prostatic Neoplasms
Keywords: Phase 1; Phase 2; metastatic castration-resistant prostate cancer; NUV-422; enzalutamide; Xtandi; CDK; CDK inhibition; CDK2/4/6
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant | interventions — enzalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b Dose Escalation (Experimental): NUV-422 will be administered orally at escalating dose levels in combination with enzalutamide until the recommended Phase 2 combination dose (RP2cD) is determined.
  160 mg enzalutamide will be administered orally daily throughout the 28-day cycles of NUV-422.
  Interventions: Drug: NUV-422; Drug: Enzalutamide
- Phase 2 (Experimental): NUV-422 will be administered orally at the RP2cD in combination with enzalutamide.
  160 mg enzalutamide will be administered orally daily throughout the 28-day cycles of NUV-422.
  Interventions: Drug: NUV-422; Drug: Enzalutamide

INTERVENTIONS:
Drug: NUV-422 — NUV-422 is an investigational drug for oral dosing.
Drug: Enzalutamide — Enzalutamide
  Other Names: Xtandi

SUMMARY:
NUV-422-04 is an open-label Phase 1b/2 dose escalation and expansion study designed to evaluate the safety and efficacy of NUV-422 in combination with enzalutamide. The study population is comprised of adults with mCRPC. Patients will self-administer NUV-422 and 160 mg enzalutamide orally in 28-day cycles. Patients will be treated until disease progression, toxicity, withdrawal of consent, or termination of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of metastatic castration-resistant prostate cancer with disease progression despite castrate levels of testosterone
2. Have radiographic or biochemical evidence of progression as determined by Investigator per standard criteria
3. Have no known active or symptomatic central nervous system (CNS) disease
4. Prior therapy with abiraterone required and:

   * For Phase 1b only: up to 2 prior taxane-based chemotherapy regimens allowed for castration-resistant disease
   * For Phase 2 only: Patients must not have received prior taxane-based chemotherapy for castrate-resistant disease or prior treatment with CDK inhibitors
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2
6. Adequate bone marrow and organ function
7. Eligible to receive enzalutamide
8. Life expectancy of > 6 months

Exclusion Criteria:

1. History of seizure or any condition that may predispose to seizure (prior cortical stroke or significant brain trauma)
2. Have received chemotherapy, hormonal therapy (with the exception of ongoing LHRH analogs) radiation, or biological anti-cancer therapy within 14 days prior to first dose of NUV-422 and enzalutamide
3. Received treatment with an investigational agent for any indication within 14 days for non-myelosuppressive agent or 21 days (or < 5 half-lives) for myelosuppressive agent prior to the first dose of NUV-422 and enzalutamide
4. Requires medications that are known to be strong inducers and /or inhibitors of CYP3A4/5 enzymes, except enzalutamide

   * For Phase 1b only: Requires medications that are known to be moderate inducers and /or inhibitors of CYP3A4/5 enzymes, except enzalutamide
5. Prior therapy with enzalutamide, apalutamide, darolutamide, or investigational androgen receptor inhibitors
6. Known allergy or hypersensitivity to enzalutamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Phase 1b Dose Escalation: Safety and tolerability of NUV-422 in combination with enzalutamide to determine the recommended Phase 2 combination dose (RP2cD) | During the DLT period (28 days)
  Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), dose-limiting toxicities (DLTs), and laboratory abnormalities
Phase 2 Dose Expansion: Prostate-specific antigen (PSA)-response rate (PSA-RR) | Every 4 weeks throughout study treatment, an average of 6 months
  PSA per standard criteria
Phase 2 Dose Expansion: Objective response rate (ORR) | Every 8 weeks throughout study treatment, an average of 6 months
  ORR per standard criteria

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Gabrail Cancer Center Research, Canton, Ohio
  - Pennsylvania Cancer Specialists and Research Institute, Gettysburg, Pennsylvania
  - NEXT Virginia, Fairfax, Virginia